CLINICAL TRIAL: NCT01881828
Title: A Randomized Trial of Metformin as Adjunct Therapy for Overweight Adolescents With Type 1 Diabetes
Brief Title: Metformin Therapy for Overweight Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T1DX-17-2013-506; 17-2013-506 (Other Grant/Funding Number: JDRF)
Record Dates: First submitted 2013-06-13; First posted 2013-06-20 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin 2000 mg per day
  Interventions: Drug: Metformin (glucophage)
- Oral Placebo (Placebo Comparator): A central pharmacy will compound a placebo to match the metformin tablets.
  The placebo product will contain the following components:
  * Micosolle™, silica based excipient
  * Silicified Micro Crystalline Cellulose, National Formulary
  * Safflower Oil, United States Pharmacopeia
  * K-30 Povidone Powder
  * Magnesium Stearate, National Formulary (Vegetable source)
  * Fumed Silica, National Formulary
  Interventions: Other: oral placebo

INTERVENTIONS:
Drug: Metformin (glucophage) — The strength of each tablet will be 500 mg. Participants will build up to a daily dose over four weeks by taking one tablet per day for 7 days, one tablet twice daily for 7 days, one tablet in morning and 2 tablets at night for 7 days, and then 2 tablets in the morning and 2 tablets at night, daily throughout the remainder of the study treatment period.
  Arms: Metformin
Other: oral placebo
  Arms: Oral Placebo

SUMMARY:
The objective of the proposed research is to evaluate the efficacy and safety of the use of metformin in addition to standard insulin therapy in overweight and obese children and adolescents, age 12-<20 years, with type 1 diabetes for at least 1 year. Secondary objectives are to assess the effect of metformin on C-peptide levels, a measure of how much insulin is still being produced by the beta cells of the pancreas, and on vascular dysfunction. In addition, an ancillary study is planned to assess if metformin will improve tissue-specific insulin resistance in type 1 diabetes using a hyperinsulinemic euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of presumed autoimmune type 1 diabetes (T1D) as indicated by age of diagnosis <10 years or documented positive diabetes-related autoantibodies.

   a. Note: For randomization, presence of at least one of the diabetes-related autoantibodies [Insulin autoantibodies (IAA) at diagnosis prior to initiation of insulin, Islet cell antibodies (ICA), Anti-GAD (GAD65), Anti-IA2 (IA2), Zinc Transporter 8 (ZnT8)] must be documented either from medical records or new laboratory measurement (IAA and ICA not measured by central lab) sent to central lab for participants who were ≥10 years old at diagnosis.
2. Age: 12 to <20 years.
3. Duration of type 1 diabetes: ≥1 years.
4. Current insulin regimen involves either use of an insulin pump or multiple daily injections of insulin (at least 3 shots per day) for the last three months, with no plans to switch the modality of insulin administration during the next 6 months (e.g., injection user switching to a pump, pump user switching to injections).
5. Hemoglobin A1c: 7.5% - <10.0% from point of care measurement or local lab on day of screening visit or within 1 month prior.
6. BMI: ≥85th percentile adjusted for age and sex .
7. Total daily dose of insulin: ≥0.8 units per kg per day.
8. Average of ≥3 Self-Monitoring Blood Glucose (SMBG) tests per day prior to initiating study and from download of study-provided blood glucose meter following screening visit.
9. Available for at least 6 months of follow-up, has home phone (or access to phone), and willing to be contacted by clinical site staff.
10. Expected to comply with protocol in investigator's judgment.

Exclusion Criteria:

1. Use of non-insulin medications for blood glucose control within prior 6 months or planning to use within next 6 months (other than study drug).
2. Use of medications for weight reduction (such as: Belviq (lorcaserin), Qsymia (Phentermine + topiramate), Orlistat (xenical)) within the prior 6 months or planning to use within next 6 months.
3. Use of a medication such as stimulants, psychotropic agents and oral/inhaled glucocorticoids that could affect weight gain or glycemic control of T1D or planning to use within the next 6 months.
4. Any condition that in the judgment of the investigator will adversely affect the completion of the protocol.
5. Females: pregnant, lactating, or intending to become pregnant within the next 34 weeks

   * A negative urine pregnancy test will be required for all females An effective contraceptive method or abstinence will be required for all females who have experienced menarche
   * Requirements regarding pregnancy testing prior to enrollment and monitoring for pregnancy over the course of the study may be further defined by each individual Institutional Review Board (IRB)
6. Clinical diagnosis of celiac disease that is in poor control as defined by most recent tissue transglutaminase (tTG) that is in the abnormal range.
7. History of ≥1 diabetic ketoacidosis events in the past 3 months.
8. History of ≥1 severe hypoglycemic events (cognitive impairment that required assistance to treat) in the past 3 months.
9. History of anemia or vitamin B12 deficiency in the past 2 years.
10. Participation in an intervention study in the past 3 months.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kellee Miller, MPH, Principal Investigator — Jaeb Center for Health Research; Ingrid Libman, MD, PhD, Study Chair — Childrens Hospital of University of Pittsburgh Medical Center; Kristen Nadeau, MD, Study Chair — University of Colorado Denver/Childrens Hospital Colorado
Locations (1):
- Jaeb Center for Health Research, Tampa, Florida, United States

REFERENCES:
- [Background] Libman IM, Pietropaolo M, Arslanian SA, LaPorte RE, Becker DJ. Changing prevalence of overweight children and adolescents at onset of insulin-treated diabetes. Diabetes Care. 2003 Oct;26(10):2871-5. doi: 10.2337/diacare.26.10.2871. PMID 14514594
- [Background] Kaminski BM, Klingensmith GJ, Beck RW, Tamborlane WV, Lee J, Hassan K, Schatz D, Kollman C, Redondo MJ; Pediatric Diabetes Consortium. Body mass index at the time of diagnosis of autoimmune type 1 diabetes in children. J Pediatr. 2013 Apr;162(4):736-740.e1. doi: 10.1016/j.jpeds.2012.09.017. Epub 2012 Oct 23. PMID 23092524
- [Background] Liu LL, Lawrence JM, Davis C, Liese AD, Pettitt DJ, Pihoker C, Dabelea D, Hamman R, Waitzfelder B, Kahn HS; SEARCH for Diabetes in Youth Study Group. Prevalence of overweight and obesity in youth with diabetes in USA: the SEARCH for Diabetes in Youth study. Pediatr Diabetes. 2010 Feb;11(1):4-11. doi: 10.1111/j.1399-5448.2009.00519.x. Epub 2009 May 15. PMID 19473302
- [Background] Valerio G, Iafusco D, Zucchini S, Maffeis C; Study-Group on Diabetes of Italian Society of Pediatric Endocrinology and Diabetology (ISPED). Abdominal adiposity and cardiovascular risk factors in adolescents with type 1 diabetes. Diabetes Res Clin Pract. 2012 Jul;97(1):99-104. doi: 10.1016/j.diabres.2012.01.022. Epub 2012 Feb 13. PMID 22336634
- [Background] Purnell JQ, Hokanson JE, Marcovina SM, Steffes MW, Cleary PA, Brunzell JD. Effect of excessive weight gain with intensive therapy of type 1 diabetes on lipid levels and blood pressure: results from the DCCT. Diabetes Control and Complications Trial. JAMA. 1998 Jul 8;280(2):140-6. doi: 10.1001/jama.280.2.140. PMID 9669786
- [Background] Rodriguez BL, Dabelea D, Liese AD, Fujimoto W, Waitzfelder B, Liu L, Bell R, Talton J, Snively BM, Kershnar A, Urbina E, Daniels S, Imperatore G; SEARCH Study Group. Prevalence and correlates of elevated blood pressure in youth with diabetes mellitus: the SEARCH for diabetes in youth study. J Pediatr. 2010 Aug;157(2):245-251.e1. doi: 10.1016/j.jpeds.2010.02.021. Epub 2010 Apr 14. PMID 20394942
- [Background] Nadeau KJ, Regensteiner JG, Bauer TA, Brown MS, Dorosz JL, Hull A, Zeitler P, Draznin B, Reusch JE. Insulin resistance in adolescents with type 1 diabetes and its relationship to cardiovascular function. J Clin Endocrinol Metab. 2010 Feb;95(2):513-21. doi: 10.1210/jc.2009-1756. Epub 2009 Nov 13. PMID 19915016
- [Background] Snell-Bergeon JK, Hokanson JE, Jensen L, MacKenzie T, Kinney G, Dabelea D, Eckel RH, Ehrlich J, Garg S, Rewers M. Progression of coronary artery calcification in type 1 diabetes: the importance of glycemic control. Diabetes Care. 2003 Oct;26(10):2923-8. doi: 10.2337/diacare.26.10.2923. PMID 14514603
- [Background] Chait A, Bornfeldt KE. Diabetes and atherosclerosis: is there a role for hyperglycemia? J Lipid Res. 2009 Apr;50 Suppl(Suppl):S335-9. doi: 10.1194/jlr.R800059-JLR200. Epub 2008 Nov 23. PMID 19029122
- [Background] Maahs DM, Kinney GL, Wadwa P, Snell-Bergeon JK, Dabelea D, Hokanson J, Ehrlich J, Garg S, Eckel RH, Rewers MJ. Hypertension prevalence, awareness, treatment, and control in an adult type 1 diabetes population and a comparable general population. Diabetes Care. 2005 Feb;28(2):301-6. doi: 10.2337/diacare.28.2.301. PMID 15677783
- [Background] Wadwa RP, Kinney GL, Maahs DM, Snell-Bergeon J, Hokanson JE, Garg SK, Eckel RH, Rewers M. Awareness and treatment of dyslipidemia in young adults with type 1 diabetes. Diabetes Care. 2005 May;28(5):1051-6. doi: 10.2337/diacare.28.5.1051. PMID 15855566
- [Background] Borch-Johnsen K, Kreiner S. Proteinuria: value as predictor of cardiovascular mortality in insulin dependent diabetes mellitus. Br Med J (Clin Res Ed). 1987 Jun 27;294(6588):1651-4. doi: 10.1136/bmj.294.6588.1651. PMID 3113569
- [Background] Krolewski AS, Kosinski EJ, Warram JH, Leland OS, Busick EJ, Asmal AC, Rand LI, Christlieb AR, Bradley RF, Kahn CR. Magnitude and determinants of coronary artery disease in juvenile-onset, insulin-dependent diabetes mellitus. Am J Cardiol. 1987 Apr 1;59(8):750-5. doi: 10.1016/0002-9149(87)91086-1. PMID 3825934
- [Background] Snell-Bergeon JK, Hokanson JE, Kinney GL, Dabelea D, Ehrlich J, Eckel RH, Ogden L, Rewers M. Measurement of abdominal fat by CT compared to waist circumference and BMI in explaining the presence of coronary calcium. Int J Obes Relat Metab Disord. 2004 Dec;28(12):1594-9. doi: 10.1038/sj.ijo.0802796. PMID 15467773
- [Background] Maahs DM, Ogden LG, Kinney GL, Wadwa P, Snell-Bergeon JK, Dabelea D, Hokanson JE, Ehrlich J, Eckel RH, Rewers M. Low plasma adiponectin levels predict progression of coronary artery calcification. Circulation. 2005 Feb 15;111(6):747-53. doi: 10.1161/01.CIR.0000155251.03724.A5. Epub 2005 Feb 7. PMID 15699257
- [Background] Orchard TJ, Olson JC, Erbey JR, Williams K, Forrest KY, Smithline Kinder L, Ellis D, Becker DJ. Insulin resistance-related factors, but not glycemia, predict coronary artery disease in type 1 diabetes: 10-year follow-up data from the Pittsburgh Epidemiology of Diabetes Complications Study. Diabetes Care. 2003 May;26(5):1374-9. doi: 10.2337/diacare.26.5.1374. PMID 12716791
- [Background] Libby P, Nathan DM, Abraham K, Brunzell JD, Fradkin JE, Haffner SM, Hsueh W, Rewers M, Roberts BT, Savage PJ, Skarlatos S, Wassef M, Rabadan-Diehl C; National Heart, Lung, and Blood Institute; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Report of the National Heart, Lung, and Blood Institute-National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Circulation. 2005 Jun 28;111(25):3489-93. doi: 10.1161/CIRCULATIONAHA.104.529651. No abstract available. PMID 15983263
- [Background] Lloyd CE, Kuller LH, Ellis D, Becker DJ, Wing RR, Orchard TJ. Coronary artery disease in IDDM. Gender differences in risk factors but not risk. Arterioscler Thromb Vasc Biol. 1996 Jun;16(6):720-6. doi: 10.1161/01.atv.16.6.720. PMID 8640398
- [Background] Soedamah-Muthu SS, Chaturvedi N, Toeller M, Ferriss B, Reboldi P, Michel G, Manes C, Fuller JH; EURODIAB Prospective Complications Study Group. Risk factors for coronary heart disease in type 1 diabetic patients in Europe: the EURODIAB Prospective Complications Study. Diabetes Care. 2004 Feb;27(2):530-7. doi: 10.2337/diacare.27.2.530. PMID 14747240
- [Background] Amiel SA, Sherwin RS, Simonson DC, Lauritano AA, Tamborlane WV. Impaired insulin action in puberty. A contributing factor to poor glycemic control in adolescents with diabetes. N Engl J Med. 1986 Jul 24;315(4):215-9. doi: 10.1056/NEJM198607243150402. PMID 3523245
- [Background] Arslanian S, Heil BV, Kalhan SC. Hepatic insulin action in adolescents with insulin-dependent diabetes mellitus: relationship with long-term glycemic control. Metabolism. 1993 Mar;42(3):283-90. doi: 10.1016/0026-0495(93)90075-y. PMID 8487645
- [Background] Heptulla RA, Stewart A, Enocksson S, Rife F, Ma TY, Sherwin RS, Tamborlane WV, Caprio S. In situ evidence that peripheral insulin resistance in adolescents with poorly controlled type 1 diabetes is associated with impaired suppression of lipolysis: a microdialysis study. Pediatr Res. 2003 May;53(5):830-5. doi: 10.1203/01.PDR.0000059552.08913.B7. PMID 12702748
- [Background] Hiatt WR, Huang SY, Regensteiner JG, Micco AJ, Ishimoto G, Manco-Johnson M, Drose J, Reeves JT. Venous occlusion plethysmography reduces arterial diameter and flow velocity. J Appl Physiol (1985). 1989 May;66(5):2239-44. doi: 10.1152/jappl.1989.66.5.2239. PMID 2745287
- [Background] Regensteiner JG, Popylisen S, Bauer TA, Lindenfeld J, Gill E, Smith S, Oliver-Pickett CK, Reusch JE, Weil JV. Oral L-arginine and vitamins E and C improve endothelial function in women with type 2 diabetes. Vasc Med. 2003;8(3):169-75. doi: 10.1191/1358863x03vm489oa. PMID 14989557
- [Background] Urbina EM, Wadwa RP, Davis C, Snively BM, Dolan LM, Daniels SR, Hamman RF, Dabelea D. Prevalence of increased arterial stiffness in children with type 1 diabetes mellitus differs by measurement site and sex: the SEARCH for Diabetes in Youth Study. J Pediatr. 2010 May;156(5):731-7, 737.e1. doi: 10.1016/j.jpeds.2009.11.011. Epub 2010 Jan 25. PMID 20097360
- [Background] Wadwa RP, Urbina EM, Anderson AM, Hamman RF, Dolan LM, Rodriguez BL, Daniels SR, Dabelea D; SEARCH Study Group. Measures of arterial stiffness in youth with type 1 and type 2 diabetes: the SEARCH for diabetes in youth study. Diabetes Care. 2010 Apr;33(4):881-6. doi: 10.2337/dc09-0747. Epub 2010 Jan 12. PMID 20067960
- [Background] Haller MJ, Stein J, Shuster J, Theriaque D, Silverstein J, Schatz DA, Earing MG, Lerman A, Mahmud FH. Peripheral artery tonometry demonstrates altered endothelial function in children with type 1 diabetes. Pediatr Diabetes. 2007 Aug;8(4):193-8. doi: 10.1111/j.1399-5448.2007.00246.x. PMID 17659060
- [Background] Mortensen HB, Robertson KJ, Aanstoot HJ, Danne T, Holl RW, Hougaard P, Atchison JA, Chiarelli F, Daneman D, Dinesen B, Dorchy H, Garandeau P, Greene S, Hoey H, Kaprio EA, Kocova M, Martul P, Matsuura N, Schoenle EJ, Sovik O, Swift PG, Tsou RM, Vanelli M, Aman J. Insulin management and metabolic control of type 1 diabetes mellitus in childhood and adolescence in 18 countries. Hvidore Study Group on Childhood Diabetes. Diabet Med. 1998 Sep;15(9):752-9. doi: 10.1002/(SICI)1096-9136(199809)15:93.0.CO;2-W. PMID 9737804
- [Background] Hamilton J, Cummings E, Zdravkovic V, Finegood D, Daneman D. Metformin as an adjunct therapy in adolescents with type 1 diabetes and insulin resistance: a randomized controlled trial. Diabetes Care. 2003 Jan;26(1):138-43. doi: 10.2337/diacare.26.1.138. PMID 12502670
- [Background] Cusi D, Bianchi G. A primer on the genetics of hypertension. Kidney Int. 1998 Aug;54(2):328-42. doi: 10.1046/j.1523-1755.1998.00007.x. No abstract available. PMID 9690199
- [Background] Ibanez L, Lopez-Bermejo A, Diaz M, Marcos MV, de Zegher F. Early metformin therapy (age 8-12 years) in girls with precocious pubarche to reduce hirsutism, androgen excess, and oligomenorrhea in adolescence. J Clin Endocrinol Metab. 2011 Aug;96(8):E1262-7. doi: 10.1210/jc.2011-0555. Epub 2011 Jun 1. PMID 21632811
- [Background] Kendall D, Vail A, Amin R, Barrett T, Dimitri P, Ivison F, Kibirige M, Mathew V, Matyka K, McGovern A, Stirling H, Tetlow L, Wales J, Wright N, Clayton P, Hall C. Metformin in obese children and adolescents: the MOCA trial. J Clin Endocrinol Metab. 2013 Jan;98(1):322-9. doi: 10.1210/jc.2012-2710. Epub 2012 Nov 21. PMID 23175691
- [Background] Tarkun I, Dikmen E, Cetinarslan B, Canturk Z. Impact of treatment with metformin on adipokines in patients with polycystic ovary syndrome. Eur Cytokine Netw. 2010 Dec;21(4):272-7. doi: 10.1684/ecn.2010.0217. Epub 2010 Dec 3. PMID 21126943
- [Background] Steinberg HO, Baron AD. Vascular function, insulin resistance and fatty acids. Diabetologia. 2002 May;45(5):623-34. doi: 10.1007/s00125-002-0800-2. Epub 2002 Apr 4. PMID 12107742
- [Background] Regensteiner JG, Bauer TA, Reusch JE. Rosiglitazone improves exercise capacity in individuals with type 2 diabetes. Diabetes Care. 2005 Dec;28(12):2877-83. doi: 10.2337/diacare.28.12.2877. PMID 16306548
- [Background] Agarwal N, Rice SP, Bolusani H, Luzio SD, Dunseath G, Ludgate M, Rees DA. Metformin reduces arterial stiffness and improves endothelial function in young women with polycystic ovary syndrome: a randomized, placebo-controlled, crossover trial. J Clin Endocrinol Metab. 2010 Feb;95(2):722-30. doi: 10.1210/jc.2009-1985. Epub 2009 Dec 8. PMID 19996308
- [Background] Montanari G, Bondioli A, Rizzato G, Puttini M, Tremoli E, Mussoni L, Mannucci L, Pazzucconi F, Sirtori CR. Treatment with low dose metformin in patients with peripheral vascular disease. Pharmacol Res. 1992 Jan;25(1):63-73. doi: 10.1016/s1043-6618(05)80065-9. PMID 1738759
- [Background] Pitocco D, Zaccardi F, Tarzia P, Milo M, Scavone G, Rizzo P, Pagliaccia F, Nerla R, Di Franco A, Manto A, Rocca B, Lanza GA, Crea F, Ghirlanda G. Metformin improves endothelial function in type 1 diabetic subjects: a pilot, placebo-controlled randomized study. Diabetes Obes Metab. 2013 May;15(5):427-31. doi: 10.1111/dom.12041. Epub 2012 Dec 5. PMID 23167274
- [Background] Bailey CJ. Metformin: a multitasking medication. Diab Vasc Dis Res. 2008 Sep;5(3):156. doi: 10.3132/dvdr.2008.026. No abstract available. PMID 18777487
- [Background] Liebson PR. Diabetes control and cardiovascular risk, Part II: Intensive glucose control--UKPDS follow-up. Prev Cardiol. 2009 Winter;12(1):51-8. doi: 10.1111/j.1751-7141.2008.00020.x. No abstract available. PMID 19301692
- [Background] Vella S, Buetow L, Royle P, Livingstone S, Colhoun HM, Petrie JR. The use of metformin in type 1 diabetes: a systematic review of efficacy. Diabetologia. 2010 May;53(5):809-20. doi: 10.1007/s00125-009-1636-9. Epub 2010 Jan 8. PMID 20057994
- [Background] Sarnblad S, Kroon M, Aman J. Metformin as additional therapy in adolescents with poorly controlled type 1 diabetes: randomised placebo-controlled trial with aspects on insulin sensitivity. Eur J Endocrinol. 2003 Oct;149(4):323-9. doi: 10.1530/eje.0.1490323. PMID 14514347
- [Background] TODAY Study Group; Zeitler P, Hirst K, Pyle L, Linder B, Copeland K, Arslanian S, Cuttler L, Nathan DM, Tollefsen S, Wilfley D, Kaufman F. A clinical trial to maintain glycemic control in youth with type 2 diabetes. N Engl J Med. 2012 Jun 14;366(24):2247-56. doi: 10.1056/NEJMoa1109333. Epub 2012 Apr 29. PMID 22540912
- [Background] Reinstatler L, Qi YP, Williamson RS, Garn JV, Oakley GP Jr. Association of biochemical B(1)(2) deficiency with metformin therapy and vitamin B(1)(2) supplements: the National Health and Nutrition Examination Survey, 1999-2006. Diabetes Care. 2012 Feb;35(2):327-33. doi: 10.2337/dc11-1582. Epub 2011 Dec 16. PMID 22179958
- [Background] Nadeau KJ, Ehlers LB, Zeitler PS, Love-Osborne K. Treatment of non-alcoholic fatty liver disease with metformin versus lifestyle intervention in insulin-resistant adolescents. Pediatr Diabetes. 2009 Feb;10(1):5-13. doi: 10.1111/j.1399-5448.2008.00450.x. Epub 2008 Aug 20. PMID 18721166
- [Background] Salpeter SR, Greyber E, Pasternak GA, Salpeter EE. Risk of fatal and nonfatal lactic acidosis with metformin use in type 2 diabetes mellitus. Cochrane Database Syst Rev. 2010 Apr 14;2010(4):CD002967. doi: 10.1002/14651858.CD002967.pub4. PMID 20393934
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236
- [Background] Dabelea D, D'Agostino RB Jr, Mason CC, West N, Hamman RF, Mayer-Davis EJ, Maahs D, Klingensmith G, Knowler WC, Nadeau K. Development, validation and use of an insulin sensitivity score in youths with diabetes: the SEARCH for Diabetes in Youth study. Diabetologia. 2011 Jan;54(1):78-86. doi: 10.1007/s00125-010-1911-9. Epub 2010 Oct 1. PMID 20886205
- [Derived] Libman IM, Miller KM, DiMeglio LA, Bethin KE, Katz ML, Shah A, Simmons JH, Haller MJ, Raman S, Tamborlane WV, Coffey JK, Saenz AM, Beck RW, Nadeau KJ; T1D Exchange Clinic Network Metformin RCT Study Group. Effect of Metformin Added to Insulin on Glycemic Control Among Overweight/Obese Adolescents With Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2015 Dec 1;314(21):2241-50. doi: 10.1001/jama.2015.16174. PMID 26624824

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Placebo: A central pharmacy will compound a placebo to match the metformin tablets.
  The placebo product will contain the following components:
  * Micosolle™, silica based excipient
  * Silicified Micro Crystalline Cellulose, National Formulary
  * Safflower Oil, United States Pharmacopeia
  * K-30 Povidone Powder
  * Magnesium Stearate, National Formulary (Vegetable source)
  * Fumed Silica, National Formulary
  oral placebo
Period: Overall Study
Arm/Group | Metformin | Oral Placebo
Started | 71 (23 excluded at randomization from enrollment) | 69 (23 excluded from randomization from enrollment)
Completed | 71 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Oral Placebo | Total
Number analyzed (Participants) | 71 | 69 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.7) | 15.1 (1.8) | 15.3 (1.7)
Age, Customized [Number; unit: years]
  12-15 years | 43 | 47 | 90
  16-19 years | 28 | 22 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 92
  Male | 27 | 21 | 48
Race/Ethnicity, Customized [Number; unit: participants]
  White | 51 | 52 | 103
  Black | 4 | 5 | 9
  Hispanic or Latino | 13 | 11 | 24
  Asian | 2 | 0 | 2
  More than one race | 1 | 1 | 2
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 7.5 (3.6) | 6.4 (3.0) | 7.0 (3.6)
Duration of Diabetes (group) [Number; unit: years]
  1-2 Years | 5 | 9 | 14
  3-5 Years | 23 | 25 | 48
  6-8 Years | 19 | 22 | 41
  ≥ 9 years | 24 | 13 | 37
Body Mass Index (BMI) Z Score [Mean (Standard Deviation); unit: Z score] — Body mass index z-scores are measures of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate BMI values lower than the mean and positive numbers indicate BMI values higher than the mean.
  Z score | 1.6 (0.4) | 1.7 (0.3) | 1.6 (0.3)
Body Mass Index (BMI) Percentile Group [Number; unit: participants]
  Overweight: 85th-<95th% | 36 | 26 | 62
  Obese: ≥ 95th % | 33 | 41 | 74
Tanner Staging (Pubic Hair) [Number; unit: participants] — For all three sites of development, Tanner Stage 1 corresponds to the pre-pubertal form with progression to Tanner Stage 5, the final adult form.
  participants
    Stage 1 | 1 | 1 | 2
    Stage 2 | 1 | 3 | 4
    Stage 3 | 5 | 7 | 12
    Stage 4 | 16 | 9 | 25
    Stage 5 | 48 | 49 | 97
Tanner Staging (Breasts/Genitals) [Number; unit: participants] — For all three sites of development, Tanner Stage 1 corresponds to the pre-pubertal form with progression to Tanner Stage 5, the final adult form.
  participants
    Stage 1 | 1 | 1 | 2
    Stage 2 | 0 | 2 | 2
    Stage 3 | 5 | 6 | 11
    Stage 4 | 12 | 9 | 21
    Stage 5 | 53 | 51 | 104
Highest Parent Educaiton Level [Number; unit: participants]
  High school diploma, GED, or less | 22 | 20 | 42
  Associate | 10 | 12 | 22
  Bachelor | 18 | 15 | 33
  Master | 12 | 13 | 25
  Professional | 5 | 7 | 12
  Unknown / Do not want to answer | 4 | 2 | 6
Income Category [Number; unit: participants]
  Less than $35,000 | 5 | 7 | 12
  $35,000 to less than $50,000 | 3 | 7 | 10
  $50,000 to less than $75,000 | 10 | 13 | 23
  $75,000 to less than $100,000 | 14 | 12 | 26
  $100,000 to less than $200,000 | 5 | 6 | 11
  Unknown / Do not want to answer | 23 | 18 | 41
Insurance [Number; unit: participants]
  Private Insurance | 53 | 48 | 101
  Other Insurance | 14 | 15 | 29
  None | 0 | 2 | 2
  Unknown / Do not want to answer | 4 | 4 | 8
Severe Hypoglycemia Events Since T1D Diagnosis [Number; unit: episodes]
  None | 52 | 52 | 104
  1-2 episodes | 14 | 10 | 24
  3-4 episodes | 3 | 2 | 5
  ≥ 5 episodes | 2 | 5 | 7
Diabetic Ketoacidosis Events Since T1D Diagnosis [Number; unit: episodes]
  None | 53 | 48 | 101
  1-2 episodes | 15 | 13 | 28
  3-4 episodes | 2 | 6 | 8
  ≥ 5 episodes | 1 | 2 | 3
HbA1c Lab [Mean (Standard Deviation); unit: percentage] | 8.8 (0.8) | 8.8 (0.7) | 8.8 (0.7)
HbA1c Group [Number; unit: participants]
  < 8.5% | 25 | 24 | 49
  8.5%-9.4% | 32 | 26 | 58
  ≥ 9.5% | 14 | 19 | 33
Mean Sensor Glucose [Mean (Standard Deviation); unit: mg/dL] | 206 (35) | 208 (34) | 207 (34.6)
Insulin Pump Use [Number; unit: participants] | 50 | 49 | 99
Continuous Glucose Monitor Use [Number; unit: participants] | 2 | 2 | 4
Self-Monitoring of Blood Glucose per day [Mean (Standard Deviation); unit: number of checks per day] | 4.5 (1.2) | 4.6 (1.6) | 4.5 (1.4)
Self-Monitoring of Blood Glucose group [Number; unit: participants]
  3 | 13 | 14 | 27
  4-5 | 44 | 43 | 87
  ≥ 6 | 14 | 12 | 26
Total Daily Insulin [Mean (Standard Deviation); unit: unit/kg/day] | 1.1 (0.2) | 1.1 (0.2) | 1.1 (0.2)
Total Daily Insulin Group [Number; unit: participants]
  <1.0 | 33 | 26 | 59
  1.0-1.4 | 33 | 39 | 72
  ≥ 1.5 | 5 | 4 | 9
Total Basal/Long Acting Insulin [Mean (Standard Deviation); unit: unit/kg/day] | 0.5 (0.1) | 0.5 (0.1) | 0.5 (0.1)
Body Mass Index (BMI) Percentile [Mean (Standard Deviation); unit: percentile] | 93.7 (4.1) | 94.3 (3.8) | 94 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c From Baseline to 26 Weeks, Adjusted for Baseline Hemoglobin A1c.
Description: Hemoglobin A1c is a measure of glycemic control over approximately the past 3 months
Time Frame: 0-26 weeks
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Metformin | Oral Placebo
Number analyzed (Participants) | 71 | 69
percentage
  HbA1c | 9.0 [8.8 to 9.2] | 8.9 [8.7 to 9.2]
  Change from Baseline to 26 Weeks | 0.2 [0.0 to 0.4] | 0.2 [-0.1 to 0.4]

2. Primary Outcome: Change in Hemoglobin A1c From Baseline to 26 Weeks, Adjusted for Baseline Hemoglobin A1c.
Description: Hemoglobin A1c is a measure of glycemic control over approximately the past 3 months
Time Frame: 0-26 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Metformin | Oral Placebo
Number analyzed (Participants) | 71 | 69
percentage of participants
  HbA1c Decrease ≥0.5% | 19 | 18
  HbA1c Increase ≥0.5% | 44 | 35
  HbA1c <7.5% | 3 | 4

3. Secondary Outcome: Change in Total Daily Dose of Insulin (TDI) Per kg
Time Frame: 0-26 weeks
Measure: Mean (95% Confidence Interval); unit: insulin per kg
Arm/Group | Metformin | Oral Placebo
Number analyzed (Participants) | 71 | 69
insulin per kg | -0.1 [-0.1 to -0.1] | -0.0 [-0.1 to -0.0]

4. Secondary Outcome: Change in Body Mass Index (BMI)
Time Frame: 0-26 weeks
Measure: Mean (95% Confidence Interval); unit: percentile
Arm/Group | Metformin | Oral Placebo
Number analyzed (Participants) | 71 | 69
percentile | -1 [-2 to 0] | 1 [-0.0 to 1]

5. Secondary Outcome: Change in Waist Circumference
Time Frame: 0-26 weeks
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Metformin | Oral Placebo
Number analyzed (Participants) | 71 | 69
centimeters | -0 [-2 to 1] | 1 [-1 to 3]

6. Secondary Outcome: Change in Body Composition
Description: Change in percent body fat
Time Frame: 0-26 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Metformin | Oral Placebo
Number analyzed (Participants) | 71 | 69
percentage of change | -0 [-1 to 1] | 1 [0 to 1]

7. Secondary Outcome: Change in Serum Lipids
Time Frame: 0-26 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Metformin | Oral Placebo
Number analyzed (Participants) | 71 | 69
mg/dL
  Change in LDL | -6 [-11 to -0] | 2 [-3 to 7]
  Change in VLDL | -0 [-3 to 2] | 1 [-1 to 3]
  Change in HDL | -0 [-2 to 2] | -1 [-2 to 1]
  Change in Triglycerides | 4 [-5 to 13] | 6 [-5 to 17]
  Change in Total Cholesterol | -5 [-11 to 1] | 3 [-3 to 8]

8. Secondary Outcome: Change in Blood Pressure
Time Frame: 0-26 weeks
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Metformin | Oral Placebo
Number analyzed (Participants) | 71 | 69
mm Hg
  Change in Systolic | 0 [-0 to 0] | -0 [-0 to 0]
  Change in Diastolic | 0 [-0 to 0] | 0 [-0 to 0]

9. Other Pre Specified Outcome: Change in Liver Enzymes and Serum Creatinine
Time Frame: 0-26 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Frequency of Severe Hypoglycemia
Time Frame: 26 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Frequency of Diabetic Ketoacidosis
Time Frame: 26 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Frequency of Gastrointestinal Side-effects Including Stomach Discomfort, Diarrhea, Nausea/Vomiting, Indigestion, Flatulence.
Time Frame: 26 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Frequency of Lactic Acidosis
Time Frame: 26 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Adipocytokines
Time Frame: 0-26 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Androgen Levels in Females
Time Frame: 0-26 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in C-peptide
Description: Measured with mixed meal tolerance test among participants with evidence of residual C-peptide on a non-fasting C-peptide at screening
Time Frame: 0-26-weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Vascular Dysfunction
Time Frame: 0-26 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Metformin | Oral Placebo
Serious Adverse Events (participants affected / at risk) | 3/71 | 3/69
Other Adverse Events (participants affected / at risk) | 0/71 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=71) | Oral Placebo (N=69)
Diabetic Ketoacidosis (Endocrine disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No